CLINICAL TRIAL: NCT04928222
Title: A Trial to Evaluate Placebo Microneedle Arrays in Healthy Human Volunteers (Part I), Followed by Proof of Concept Testing of Efficacy and Safety of Doxorubicin Microneedle Arrays in Subjects With Basal Cell Cancer (Part II)
Brief Title: Placebo Microneedles in Healthy Volunteers (Part I) and Efficacy/Safety of Doxorubicin Microneedles in Basal Cell Cancer Subjects (Part II)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SkinJect, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKNJCT-002
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Neoplasms, Basal Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigational product will have randomly generated product code on label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Doxorubicin-containing MNA - 100 µg (Active Comparator): A doxorubicin-containing array of 100 µg will be applied to subjects.
  Interventions: Combination Product: Doxorubicin-containing MNA
- Placebo MNA for Training (Experimental): Training phase for application of arrays
  Interventions: Drug: Placebo-containing MNA

INTERVENTIONS:
Combination Product: Doxorubicin-containing MNA — A 15 x 15 millimeter array containing 400 dissolvable microneedles delivering active agent
  Arms: Doxorubicin-containing MNA - 100 µg
Drug: Placebo-containing MNA — A 15 15 x 15 millimeter array containing 400 dissolvable microneedles containing placebo
  Arms: Placebo MNA for Training

SUMMARY:
Part I is designed as a study of P-MNA application in healthy human volunteers. The goal of Part I is to determine several factors possibly affecting the rate and extent of microneedle array dissolution, such as anatomic location; age; duration of array exposure to the skin; and the criticality of proper array application to the skin. Part II will be a randomized study in which doxorubicin-containing arrays will be applied to subjects demonstrated by biopsy to have basal cell cancer. A subject will be randomized to one of four dose groups: placebo microneedle array and 50 µg, 100 µg, and 200 µg doses of doxorubicin in a tip-loaded, dissolvable microneedle arrays (D-MNA).

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, 18+ years in general good health as assessed by the investigator.
2. Clinical laboratory results within the following ranges:

   1. granulocytes ≥2,000/mm3
   2. platelets >50,000/mm3
   3. serum creatinine ≤2X the upper limit of normal (ULN)
   4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), lactate dehydrogenase (LDH), alkaline phosphatase ≤3X the ULN.
3. Subject must have no other "clinically significant" abnormal findings in his/her medical history, physical examination or clinical laboratory test results as assessed by the investigator.
4. Subject must be willing to adhere to the instructions of the investigator and his or her research team.
5. Subject must sign an Informed Consent Form prior to any study specific procedures and entry into the study.
6. BCC (subtype: superficial or nodular) confirmed histologically by diagnostic shave biopsy at the Screening Visit. If previously confirmed, subjects can only have diagnosed BCC via shaved biopsy within 6 months of first study treatment.
7. Biopsy removed ≤25% of the original volume of the target lesion.
8. Primary BCC (i.e., no previous treatment)
9. Lesion size ≥ 64 mm2 or 8 x 8 mm and ≤ 169 mm2 or 13 x 13 mm, i.e., the entire lesion must be covered by 13X13 mm area of the array containing the microneedles
10. Subjects must avoid sunlight/ultraviolet light to the target lesion for the duration of the study.
11. Female subjects must be:

    1. postmenopausal (no menstrual period for a minimum of 12 months), or
    2. surgically sterile upon entry into the study.
    3. female subjects of childbearing potential must have a negative pregnancy test upon entry into this study and agree to use a highly effective method of contraception from Screening until the final follow-up visit. Consult Section 5.5 in this protocol for a description of effective contraceptive methods. Female subjects must also have negative pregnancy tests before each dose is applied to female subjects
12. Male subjects with female partners of child bearing potential must be either surgically sterile or agree to use a double-barrier contraception method (i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam) from screening until the final follow-up visit.

Exclusion Criteria:

1. Evidence of clinically significant, unstable medical conditions as assessed by the investigator.
2. Previously demonstrated sensitivity to doxorubicin or carboxymethyl cellulose.
3. Female subjects who are pregnant or breastfeeding.
4. The subject has uncontrolled, significant intercurrent or recent illness.
5. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g. dabigatran), betrixaban, or platelet inhibitors (eg, clopidogrel). Prophylactic use of Low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH) are permitted.
6. Topical therapy(ies) to the target lesion within 6 weeks of first treatment.
7. Prior excisional surgery performed on the lesion to be treated in this study.
8. Recent therapy(ies) to the BCC treatment area.
9. Recurrent BCC (previously treated) at the site presented for treatment.
10. BCC lesion to be treated is located in an area where excisional biopsy is undesired or aesthetically unacceptable to the subject
11. Subject with other active malignancies except for non-metastatic prostate cancer, carcinoma in situ of the skin or cervix, and basal cell cancer in locations other than lesion of interest.
12. Subject with evidence of metastatic malignancies.
13. Concomitant disease requiring systemic immunosuppressive treatment.
14. Genetic skin cancer disorder, e.g., basal cell nevus syndrome.
15. Subject is currently participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment (patients who are in a follow-up phase of an investigational study may participate as long as it has been 30 days after the last dose of the previous investigational agent).
16. Evidence of dermatological disease or confounding skin condition within 3 mm margin of the target BCC lesion, e.g., SCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema.
17. Existing condition or treatment within 3 months prior to the Screening Visit that may have impact on clinical outcome for the treatment of BCC or delay in wound healing from the standard of care excision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Eradication of Basal Cell Cancer based on Histologic Analysis | Up to 4 weeks after the last array application to a subject
  Tissue will be excised and sectioned for histologic analysis
Number of subjects with dose-limiting toxicity and treatment-related adverse events by CTCAE v4.0 | Assessment at week 2 of subject visit
  Determination of cutaneous tolerability of arrays after application

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Buttler, Study Director — SkinJect, Inc.
Locations (2):
- United States (2):
  - Beer Dermatology, West Palm Beach, Florida
  - New York and Presbyterian Hospital, New York, New York